CLINICAL TRIAL: NCT06948032
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BLU-808 and to Assess the Drug-Drug Interaction With a CYP3A Substrate (Midazolam) and the Effect of Food in Healthy Adult Subjects
Brief Title: Study of BLU-808 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLU-808-0101
Record Dates: First submitted 2025-04-22; First posted 2025-04-28 (Actual); Last update posted 2025-04-28 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parts 1 and 2 are double-blind and placebo-controlled. Part 3 is open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1: BLU-808 (Experimental): BLU-808 will be administered orally.
  Interventions: Drug: BLU-808
- Part 1: Placebo (Placebo Comparator): Matching placebo for BLU-808 will be administered orally.
  Interventions: Drug: Placebo
- Part 2: BLU-808 (Experimental): BLU-808 will be administered orally.
  Interventions: Drug: BLU-808
- Part 2: Placebo (Placebo Comparator): Matching placebo for BLU-808 will be administered orally.
  Interventions: Drug: Placebo
- Part 2: Midazolam Alone Followed by BLU-808 and Midazolam (Experimental): Participants will receive oral midazolam in Period 1. Participants will then receive oral BLU-808 with midazolam in period 2.
  Interventions: Drug: BLU-808; Drug: Midazolam
- Part 2: Midazolam Alone Followed by BLU-808 Matching Placebo and Midazolam (Placebo Comparator): Participants will receive oral midazolam in Period 1. Participants will then receive oral matching placebo for BLU-808 with midazolam in period 2.
  Interventions: Drug: Placebo; Drug: Midazolam
- Part 3: BLU-808 (Treatment D, E) (Experimental): BLU-808 will be administered orally.
  Interventions: Drug: BLU-808
- Part 3: BLU-808 (Treatment E, D) (Experimental): BLU-808 will be administered orally.
  Interventions: Drug: BLU-808

INTERVENTIONS:
Drug: BLU-808 — BLU-808 will be administered per schedule specified in the arm description.
  Arms: Part 1: BLU-808; Part 2: BLU-808; Part 2: Midazolam Alone Followed by BLU-808 and Midazolam; Part 3: BLU-808 (Treatment D, E); Part 3: BLU-808 (Treatment E, D)
Drug: Placebo — BLU-808 matching placebo will be administered per schedule specified in the arm description.
  Arms: Part 1: Placebo; Part 2: Midazolam Alone Followed by BLU-808 Matching Placebo and Midazolam; Part 2: Placebo
Drug: Midazolam — Midazolam will be administered per schedule specified in the arm description.
  Arms: Part 2: Midazolam Alone Followed by BLU-808 Matching Placebo and Midazolam; Part 2: Midazolam Alone Followed by BLU-808 and Midazolam

SUMMARY:
This is a 3-part study. Parts 1 and 2 are randomized, double-blind, placebo-controlled investigations of single ascending doses (SAD) (Part 1) and multiple ascending doses (MAD) (Part 2) of orally administered BLU-808 in healthy adult participants. Part 2 will also include an evaluation of the effect of multiple doses of BLU-808 on the single-dose pharmacokinetics (PK) of midazolam. Part 3 is an open-label, 2-sequence, 2-period, food effect (FE) study in healthy adult participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the first dosing based on subject self-reporting.
* Medically healthy with no clinically significant medical history, physical examination, clinical laboratory profiles, or vital signs, as deemed by the Principal Investigator (PI) or designee.
* No clinically significant cardiac history as judged by the PI or designee at the screening visit and check-in.

Key Exclusion Criteria:

* Participant is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* Participant has history or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI, designee, or Sponsor.
* Participant has history or presence of alcohol or drug abuse within the past 2 years prior to the first dosing.
* Participant has positive results at the screening visit for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
* Participant has been on a diet incompatible with the on-study diet (that is, unusual meal habits and special diet requirements or unwillingness to eat the food provided in the trial), in the opinion of the PI or designee, within the 30 days prior to the first dosing and throughout the study.
* Participant has participated in another clinical study within 30 days prior to the first dosing. The 30-day window will be derived from the date of the last dosing in the previous study to the first dosing of the current study.
* Participant has positive coronavirus disease 2019 (COVID-19) results at first check-in.

Note: Other protocol-specified inclusion and exclusion criteria may apply.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to Day 20
Part 2: Number of Participants With TEAEs | Up to Day 50
Part 3: Area Under the Plasma Concentration-time Curve From Time 0 to the Last Measurable Non-zero Concentration (AUC0-t) | Up to Day 6
Part 3: Maximum Observed Plasma Concentration (Cmax) | Up to Day 6

SECONDARY OUTCOMES:
Part 1: AUC0-t | Up to Day 6
Part 1: Cmax | Up to Day 6
Part 1: Terminal Elimination Half-life (t1/2) | Up to Day 6
Part 1: Change From Baseline in QTc (Corrected Value of the Interval Between the Q and T Waves on the Electrocardiogram Tracing) | Up to Day 6
Parts 1 and 2: Change From Baseline in Serum Tryptase Concentrations | Up to Day 6
Part 2: AUC0-t | Up to Day 14
Part 2: Cmax | Up to Day 14
Part 2: t1/2 | Up to Day 19
Part 3: Number of Participants With TEAEs | Up to Day 26

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Inc., Lincoln, Nebraska, United States